CLINICAL TRIAL: NCT07181603
Title: Resilience Enhancement Training Program to Confront Nursing Students' Perceived Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25.04.662
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Perceived Stress
Keywords: Resilience; Perceived stress; Stress management; Nursing students; Resilience training program

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel groups: an intervention group receiving the resilience enhancement training program and a control group receiving no intervention during the study period. The control group will be offered the training after study completion to ensure fairness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - Resilience Enhancement Training Program (Experimental): Participants in this group will receive the Resilience Enhancement Training Program in addition to their usual curriculum. The program consists of 10 weekly sessions designed to improve resilience and reduce perceived stress. Sessions include self-awareness, self-regulation, stress and coping strategies, cognitive restructuring, self-compassion, gratitude practice, optimism training, self-esteem, and a wrap-up with evaluation.
  Interventions: Behavioral: Resilience Enhancement Training Program
- Control Group - Usual Curriculum (No Intervention): Participants in this group will continue with their usual nursing curriculum during the study period and will not receive the training program. To ensure fairness, the Resilience Enhancement Training Program will be offered to this group after the completion of the study.

INTERVENTIONS:
Behavioral: Resilience Enhancement Training Program — A structured 10-week behavioral training program designed to improve resilience and reduce perceived stress among nursing students. The program includes 10 sessions covering self-awareness, self-regulation, stress and coping strategies, cognitive restructuring, self-compassion, gratitude practice, optimism training, self-esteem, and a wrap-up with evaluation. Each session aims to strengthen coping skills and psychological adaptability.
  Arms: Intervention Group - Resilience Enhancement Training Program

SUMMARY:
The goal of this clinical trial is to assess if a resilience enhancement training program can help nursing students manage stress more effectively. The main question it aims to answer is:

Does the program improve nursing students' resilience levels?

Does the program lower nursing students' perceived stress levels?

Researchers will compare students who receive the training during the semester with students who do not receive it until after the study is completed to see if the training has an effect.

Participants will:

1. Complete questionnaires on resilience and stress before and after the training.
2. Attend a structured resilience enhancement training program for 10 weeks alongside their usual studies.
3. Be part of either the study group (receiving the training first) or the comparison group (receiving the training after study completion).

DETAILED DESCRIPTION:
This quasi-experimental study is designed to evaluate the effect of a resilience enhancement training program on perceived stress among nursing students. Nursing students commonly face high academic and clinical demands, long working hours, and frequent exposure to emotionally challenging situations. Such pressures often lead to elevated stress levels, anxiety, and potential burnout, which can impair learning, professional growth, and the quality of patient care. Evidence from prior studies (e.g., meta-analyses of stress-management interventions in healthcare students) indicates that programs focused on resilience building-such as cognitive restructuring, mindfulness, and self-compassion practices-can strengthen coping skills, reduce perceived stress, and enhance well-being.

Low resilience has been associated with higher susceptibility to stress and psychological distress. Interventions that explicitly teach resilience skills may empower students to adapt more effectively and sustain academic performance. Building on this evidence, the present study aims to:

1. Assess baseline resilience and perceived stress levels among nursing students.
2. Develop and implement a 10-week structured resilience enhancement training program tailored to the needs of nursing students.
3. Evaluate the impact of the program on resilience and perceived stress by comparing outcomes between a study group and a control group.

Hypothesis:

The resilience enhancement training program will significantly increase resilience levels and reduce perceived stress levels among nursing students.

Design and Methods:

A quasi-experimental research design with study and control groups will be used. Participants will be undergraduate nursing students enrolled in the Psychiatric and Mental Health Nursing (PMHN) course at the Faculty of Nursing, Ain Shams University, during the first semester of the academic year 2025-2026. Students will be randomly allocated into two groups:

Study group: Receives the resilience enhancement training program in addition to their standard curriculum.

Control group: Follows the standard curriculum during the study period and will receive the program after the study ends to ensure fairness.

Sample size: all nursing students who enrolled in the psychiatric and mental health nursing course will be included in this study. Participation will be voluntary, and written informed consent will be obtained.

Intervention Structure: The 10-week resilience enhancement training program includes structured sessions (approximately 90 minutes each) that cover key skills such as self-awareness, self-regulation, stress management, cognitive restructuring, self-compassion, gratitude practices, optimism training, and self-evaluation. Each session has a specific objective to build coping skills and strengthen resilience. The program concludes with a wrap-up and evaluation session.

Data Collection and Evaluation

Data will be collected at two time points:

* Pre-intervention: October 2025
* Post-intervention: immediately after program completion in December 2025

Outcomes:

* Primary outcome: change in perceived stress levels measured by validated stress-scale instruments.
* Secondary outcome: change in resilience scores assessed with a standardized resilience scale. Fidelity of program delivery will be monitored through attendance records and facilitator checklists.

Ethical Considerations and Significance Ethical approval was obtained from the Scientific Research Ethics Committee, Faculty of Nursing, Ain Shams University (Study Number: 25.04.662; Approval Date: March 17, 2025). Participation is voluntary, and confidentiality will be maintained.

Findings are expected to demonstrate the effectiveness of a structured resilience-enhancement training program in strengthening students' coping skills and reducing perceived stress.

The results will guide future training programs designed to help undergraduate nursing students manage stress more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students enrolled in the Psychiatric and Mental Health Nursing (PMHN) course at the Faculty of Nursing, Ain Shams University during the first semester of the academic year 2025-2026.
* Willing to participate and able to provide informed consent

Exclusion Criteria:

* Students who decline participation or withdraw consent at any time.
* Students absent for the majority of the program sessions.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-02 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Score | Baseline (October 2025) and immediately post-intervention (December 2025)
  Perceived stress will be measured using the Perceived Stress Scale. The scale consists of 29 items, each rated on a 5-point Likert scale (0 = never to 4 = very often), yielding a total score range of 0 to 116.
  Higher total scores indicate higher levels of perceived stress (worse outcome).

SECONDARY OUTCOMES:
Change in Resilience Score | Baseline (October 2025) and post-intervention (December 2025)
  Resilience will be assessed using the full Connor-Davidson Resilience Scale. This validated instrument contains 25 items, each rated on a 5-point Likert scale (0 = not true at all to 4 = true nearly all the time), giving a total score range of 0 to 100.
  Higher total scores indicate greater psychological resilience (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Amal E Nossier, PhD, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Nursing, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sheu, S., Lin, H., Hwang, S., Yu, P., Hu, W. and Lou, M. (1997) The Development and Testing of Perceived Stress Scale of Clinical Practice. Nursing Research (Republic of China), 5, 341-351.
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174